CLINICAL TRIAL: NCT02121717
Title: Phase III Study of Chiglitazar in Patients With Type 2 Diabetes Mellitus and Insufficient Glycemic Control Despite Diet and Exercise -- A Multicenter, Randomized, Double-Blind, and Placebo-Controlled Trial
Brief Title: Study of Chiglitazar Compare With Placebo in Type 2 Diabetes Patients
Acronym: CMAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CGZ301
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes
Keywords: Chiglitazar,diabetes,type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — chiglitazar; phospholamban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Patients administrate Chiglitazar 32mg once daily for 52 weeks
  Interventions: Drug: Chiglitazar
- Arm 2 (Experimental): Patients administrate Chiglitazar 48mg once daily for 52 weeks
  Interventions: Drug: Chiglitazar
- Arm 3 (Placebo Comparator): Patients administrate placebo for 24 weeks.From week 25 to 52, patients are randomly switched to Arm 1 and Arm 2, and receive the treatment accordingly.
  Interventions: Drug: Chiglitazar; Drug: Placebo

INTERVENTIONS:
Drug: Chiglitazar — Take orally
  Other Names: CS038
Drug: Placebo — Take orally
  Other Names: Plb
  Arms: Arm 3

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Chiglitazar, compare with placebo.

DETAILED DESCRIPTION:
The efficacy and safety will be compared between Chiglitazar and placebo after treatment of 24 weeks. The long term efficacy and safety of Chiglitazar will be evaluated after 52 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the WHO Diagnostic Criteria for Type 2 Diabetes (published on 1999);
2. HbA1c≥ 7.5% and ≤ 10.0% after control of diet and exercises;
3. Male and female,age between 18 and 70 years;
4. BMI between 18.5-35kg/m2;
5. Willing to be assigned to any treatment arm and sign inform consent.

Exclusion Criteria:

1. Type 1 diabetes;
2. Treated by oral or injective antidiabetic drug before screening, including insulin and herb;
3. Fasting plasma glucose > 13.3 mmol/L (240 mg/dL);
4. Resistant hypertension [blood pressure above the goal despite adherence to at least 3 optimally dosed antihypertensive medications (including diuretic) of different classes,or blood pressure is controlled to below the goal by at least 4 different classes of drugs];
5. Plasma triglyceride > 500 mg/dL (5.65 mmol/L);
6. Is treating by fibrates;
7. History of diabetic ketoacidosis,diabetic hyperglycemic hyperosmolar syndrome,lactic acidosis, diabetic hypoglycemia; or is currently combined with retinopathy, diabetic nephropathy and diabetic neuropathy;
8. Had transient ischemic attack,cerebrovascular accident or unstable angina in the past 6 months;
9. History of myocardial infarction or had conducted coronary angioplasty or coronary artery bypass graft surgery;
10. Heart failure (NYHA classification Stage III or IV), or left ventricular hypertrophy indicated by ECG;
11. Hepatic diseases such as hepatocirrhosis, active hepatitis,aspartate aminotransferase or alanine aminotransferase > 2.5 fold of the upper limit of the normal range;
12. Kidney diseases or serum creatinine exceed the normal range: male > 133 μmol/L or female >108 μmol/L;
13. Had malignancy in the past 5 years, not including basal cell carcinoma;
14. Had or is currently receiving treatment that can alter blood glucose metabolism, including but not limited to diuretic,hormone (corticotropin or steroids),beta blockers;
15. Have the diseases that can alter blood glucose metabolism, including but not limited to active hepatitis, hyperthyroidism,or adrenal tumors;
16. Edema with unknown reason;
17. Alcohol or drug addiction;
18. Had participated other drugs' clinical trials in the 3 months before screening;
19. Pregnant or lactic women; or women of childbearing age who are not able to or is not willing to conduct contraception;
20. Any condition that make investigator consider the subject is not suitable to participate the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2014-06; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline after 24 weeks of treatment | 24 weeks
  The change of HbA1c at week 24 from baseline

SECONDARY OUTCOMES:
Change in HbA1c from baseline for patients with a baseline HbA1c >=8.5% | 24 weeks
  The change of HbA1c at week 24 from baseline for patients with a HbA1c >=8.5% at baseline
Change in HbA1c from baseline in patients with a baseline HbA1c < 8.5% | 24 weeks
  The change of HbA1c at week 24 from baseline for patients with a HbA1c < 8.5% at baseline
Change in HbA1c from baseline | 12 weeks
  The change of HbA1c at week 12 from baseline
Change in HbA1c from baseline | 52 weeks
  The change of HbA1c at week 52 from baseline
Percentage of patients that attained target HbA1c <7.0% | 24 weeks
  Percentage of patients whose HbA1c at week 24 are < 7.0%
Percentage of patients whose HbA1c lowered by at least 0.5% | 24 weeks
  Percentage of patients whose change of HbA1c at week 24 from baseline are >= 0.5%
Change in fasting plasma glucose from baseline | 12,24 and 52 weeks
  The change of fasting plasma glucose at week 12 and 24 from baseline
Change in 2-h postprandial glucose (2hPPG) from baseline | 12, 24 and 52 weeks
  The change of 2-h postprandial glucose (2hPPG) at week 12, 24 and 52 from baseline
Change in total cholesterol (TC) from baseline | 12, 24 and 52 weeks
  The change of total cholesterol (TC) at week 12, 24 and 52 from baseline
Change in triglyceride from baseline | 12,24 and 52 weeks
  The change of triglyceride at week 12, 24 and 52 from baseline
Change in high density lipoprotein cholesterol (HDL-C)from baseline | 12, 24 and 52 weeks
  The change of high density lipoprotein cholesterol (HDL-C) at week week 12, 24 and 52 from baseline
Change in low density proprotein cholesterol (LDL-C) from baseline | 12, 24 and 52 weeks
  The change of low density lipoprotein cholesterol (LDL-C) at week 12, 24 and 52 from baseline
Change in free fatty acid (FFA) from baseline | 12, 24 and 52 weeks
  The change of free fatty acid (FFA) at week 12, 24 and 52 from baseline
Change in fasting plasma insulin from baseline | 12, 24 and 52 weeks
  The change of fasting plasma insulin at week 12, 24 and 52 from baseline
Insulin sensitivity assessed by the homeostatic model assessment (HOMA) at 12,24 and 52 weeks, compared with that of baseline | 12, 24 and 52 weeks
  The change of insulin sensitivity at week 12, 24 and 52 from baseline
Change in blood pressure from baseline | 24 weeks
  The change of blood pressure at week 24 from baseline
Percentage of patients who use rescue therapy | 52 weeks
  The percentage of patients who use rescue therapy during the 52 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Dr., Principal Investigator — Peking University People's Hospital
Locations (26):
- China (26):
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - China Meitan General Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The 306th Hospital of PLA, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Cangzhou's Central Hospital, Cangzhou, Hebei
  - Harrison International Peace Hospital, Hengshui, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Ha'erbin Medical University, Harbin, Heilongjiang
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - Baogang Hospital of Inner Mongilia, Baotou, Inner Mongolia
  - The people's Hospital of Jiangsu Province, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The Affiliated Hospital of Qingdao Medical University, Qingdao, Shandong
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The Central Hospital of Yangpu District of Shanghai, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of The 4th Military Medical University, Xi’an, Shanxi
  - Huaxi Hopsital of Sichuan University, Chengdu, Sichuan
  - The General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No